CLINICAL TRIAL: NCT06014385
Title: A Trial to Evaluate Target Occupancy of Scopolamine at the Muscarinic M1 Receptor
Brief Title: PET and MRI Imaging With Scopolamine at the Muscarinic M1 Receptor
Acronym: emo_to2
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Yale University (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, David Matuskey, Associate Professor, Yale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000034723; 000 (Other: CTGTY)
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2024-12

CONDITIONS: Muscarinic Receptor Occupancy
MeSH Terms: interventions — Scopolamine; LSN3172176

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Scopolamine high dose (Experimental): The target occupancy (TO) of scopolamine at M1 will be evaluated using the radiotracer [11C]EMO and positron emission tomography (PET). TO will be measured following a 15-minute IV infusion of 4.0 μg/kg scopolamine in 4-6 anticipated participants.
  Interventions: Drug: Scopolamine; Radiation: [11C]EMO ([11C]LSN3172176)
- Scopolamine low dose (Experimental): The target occupancy (TO) of scopolamine at M1 will be evaluated using the radiotracer [11C]EMO and positron emission tomography (PET). TO will be measured following a 15-minute IV infusion of 2.0 μg/kg scopolamine in 0-2 anticipated participants.
  Interventions: Drug: Scopolamine; Radiation: [11C]EMO ([11C]LSN3172176)

INTERVENTIONS:
Drug: Scopolamine — TO will be measured following a 15-minute IV infusion of up to 2 dose levels of scopolamine: 4.0 μg/kg and 2.0 μg/kg
Radiation: [11C]EMO ([11C]LSN3172176) — A radiotracer specific for imaging M1 receptors. For each PET scan, up to 20 mCi of [11C]EMO i.v. will be administered twice, at baseline and post dosing with scopolamine.

SUMMARY:
The purpose of this study is to assess the target occupancy (TO) of scopolamine at M1 Muscarinic Receptors in the brain after single I.V. doses of scopolamine, in healthy control subjects, using the radiotracer [11C]EMO (also known as [11C]LSN3172176).

DETAILED DESCRIPTION:
Each participant will complete a baseline (pre-dose) PET scan and a post-dose PET scan, following a 15-minute IV infusion of scopolamine. Each participant will also complete a magnetic resonance imaging (MRI) scan of the brain. The timing of the post scopolamine [11C] EMO PET scan tracer injection could occur 15 minutes to 48 hours after the scopolamine infusion has been completed.

In this study, the post scopolamine [11C] EMO PET scan tracer injection should be given 4 hours (± 5 minutes) after the scopolamine infusion of 4.0 μg/kg in up to 2 subjects. The data from those 2 subjects will be reviewed to determine the timepoint for tracer injection for the post scopolamine [11C] EMO PET scan in the next 2 subjects (e.g., tracer injection at 24-hour or 1-hour post-dose). If the baseline and post scopolamine PET scans are obtained on the same day, the scopolamine infusion should be started after the acquisition of the baseline PET scan has been completed. The data from the first 4 subjects will be reviewed to determine the dose level and timepoint for tracer injection in the last 2 subjects. . At least 2 hours should elapse between injections of [11C] EMO to allow for clearance of the tracer signal from the baseline scan and the injection of [11C] EMO for a post scopolamine PET scan should not be given during a scopolamine infusion. Participants will complete at least 2 visits and up to 4.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give voluntary, written informed consent
* Have the ability to read and write, communicate effectively with the investigator and to comply with all study requirements, restrictions, and directions of the research staff.
* Male or female, aged Age 18 to 60 years inclusive, at screening.
* In good general health as evidenced by medical history, physical examination, ECG, serum/urine biochemistry, hematology, and serology tests.

Exclusion Criteria:

* History or presence of clinically significant respiratory, GI, renal, hepatic, pancreatic, hematological, neurological (including history of seizure), cardiovascular, psychiatric (including known addictive disorders), musculoskeletal, genitourinary, immunological, or dermatological disorders, including all cancers.
* Laboratory tests with clinically significant abnormalities or positive urine toxicology, at screening.
* Abnormal and clinically significant ECG, as (as determined by the Investigator or his/her designee) at screening.
* Seropositive for hepatitis B, hepatitis C, and/or HIV
* Pregnancy or lactation
* Use of prescription medications within 14 days of scopolamine dosing. Exceptions may be allowed only if the medication's administration is deemed unlikely to impact the study result.
* Current or recent use (within 14 days) of scopolamine transdermal patch, for any reason (ex: for motion sickness).
* Use of drugs with anticholinergic properties within 14 days of scopolamine dosing, for example, belladonna alkaloids, first generation antihistamines, antidepressants (tricyclics and MAO inhibitors), phenothiazines and second generation antipsychotics (clozapine and olanzapine), amantadine and quinidine. Non-sedating antihistamines (e.g., loratadine) use is acceptable.
* Strong CYP3A4 inhibitors such as itraconazole and grapefruit juice should also not be taken within 14 days of receiving scopolamine. Use of CYP3A4 inducers (e.g., carbamazepine, rifampin) should not be taken within 21 days of scopolamine administration.
* Treatment with another investigational drug or other intervention within 30 days of the screening visit, or participation in another trial involving radiotracer administration within 1 week of dosing day.
* Current smoker (including any form of nicotine use)
* History of alcohol or drug abuse, within 2 years prior to screening, as determined by the investigator.
* Positive drug test at screening
* Blood donation within eight weeks of the start of the study. Subjects that confirm recent blood donation may reschedule for a later screening date.
* History of a bleeding disorder or are currently taking anticoagulants (such as Coumadin, Heparin, Pradaxa, Xarelto).
* Unable to safely discontinue or hold aspirin and other NSAID use, as outlined in Section 6.1.8
* MRI incompatible implants (i.e., such as pacemaker, artificial joints, non-removable body piercings) and other contraindications for MRI, such as claustrophobia, having implanted or embedded metal objects/fragments or fragments in the head or body that would present a risk during the MRI scanning procedure, or have worked with ferrous metals either as a vocation or hobby (for example, as a sheet metal worker, welder, or machinist).
* Participation in other research studies involving ionizing radiation within one year of the PET scans that would cause the subject to exceed the yearly dose limits for healthy volunteers set by the Yale University PET Center. This limit follows the guidelines listed in 21 CFR 361.1 for research subjects.
* Subjects with a history of IV drug use that would prevent venous access for PET tracer injection.
* Subject who has current, past, or anticipated exposure to radiation in the work place within one year of the proposed research scans that in combination with the study tracer would result in a cumulative exposure that exceeds recommended exposure limits.
* Has any condition that, in the opinion of the investigator, would prevent compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in brain muscarinic receptor occupancy with [11C]LSN3172176 PET | baseline and up to 48 hours post scopolamine infusion
  M1 Muscarinic receptor occupancy in the brain following a 15-minute IV infusion of scopolamine in healthy adult participants using PET scans.

CONTACTS AND LOCATIONS:
Overall Officials: David Matuskey, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No